CLINICAL TRIAL: NCT03250494
Title: Impact of Duloxetine and Dexamethasone for Improving Postoperative Pain After Laparoscopic Gynecological Surgeries: a Randomized Clinical Trial
Brief Title: Duloxetine and Dexamethasone for Improving Postoperative Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Dr.Ibrahim Mamdouh Esmat, Lecturer of Anesthesia and Intensive Care Department, Faculty of Medicine, Ain- shams University, Cairo, Egypt., Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 17585
Record Dates: First submitted 2017-08-11; First posted 2017-08-15 (Actual); Last update posted 2017-08-15 (Actual); Status verified 2017-08

CONDITIONS: Post Operative Pain Control
Keywords: Duloxetine, Dexamethasone, Postoperative pain, side effects.
MeSH Terms: conditions — Pain, Postoperative | interventions — Duloxetine Hydrochloride; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- group (I) (GI) (n=25) (Active Comparator)
  Interventions: Drug: Dulox capsule (60mg)
- group (II) (GII) (n=25) (Active Comparator)
  Interventions: Drug: combined Dulox capsule (60 mg) orally and Dex 0.1mg/kg diluted in 100 ml 0.9% NS IVI
- group (III) (GIII) (control group) (n=25) (Placebo Comparator)
  Interventions: Drug: a placebo capsule identical to Dulox capsule and 100 ml 0.9% NS IVI over 15 min, as a placebo for dexamethasone

INTERVENTIONS:
Drug: Dulox capsule (60mg) — each patient received Dulox capsule (60mg) orally with sips of water 2 hours preoperatively and 100 ml 0.9% sodium chloride solution (NS) intravenous infusion (IVI) over 15 min
  Other Names: Dulox was presented as CYMBALTA® capsules manufactured by Lilly del Caribe Inc.
  Arms: group (I) (GI) (n=25)
Drug: combined Dulox capsule (60 mg) orally and Dex 0.1mg/kg diluted in 100 ml 0.9% NS IVI — each patient received combined Dulox capsule (60 mg) orally with sips of water and Dex 0.1mg/kg diluted in 100 ml 0.9% NS IVI over 15 min, 2 hours preoperatively
  Other Names: Dex was presented as dexamethasone sulphate ampoules 8mg in 2ml. (Medical Union Pharmaceutical, Egypt MUP)
  Arms: group (II) (GII) (n=25)
Drug: a placebo capsule identical to Dulox capsule and 100 ml 0.9% NS IVI over 15 min, as a placebo for dexamethasone — each patient received a placebo capsule identical to Dulox capsule and 100 ml 0.9% NS IVI over 15 min, as a placebo for dexamethasone 2 hours preoperatively.
  Arms: group (III) (GIII) (control group) (n=25)

SUMMARY:
75 female patients were randomly allocated into one of three equal groups. Group I(GI) received Dulox 60 mg orally and 100 ml 0.9% sodium chloride solution (NS) intravenous infusion (IVI) over 15 min, group II(GII): received combined Dulox capsule 60 mg orally and Dex 0.1mg/kg mixed with 100 ml NS IVI and group III(GIII) received identical placebo duloxetine capsule and 100 ml NS IVI as a placebo for Dex, 2 hours preoperatively. Patients' vitals, VAS and sedation score were assessed at 30 minutes, 1h, 2 h, 6h and 12h postoperatively. Total pethidine requirements, plasma cortisol, PONV and patient's satisfaction were recorded.

DETAILED DESCRIPTION:
This study was designed to be a randomized, placebo-controlled, double-blinded parallel study and this study was carried out at Ain-Shams university hospitals, from December 2014 to January2016, on 75 female patients aged between 25 and 35 years old of the American Society of Anesthesiologists (ASA) physical status I and II scheduled for elective laparoscopic gynecological surgeries (for infertility) under general anesthesia. Approval was obtained from the institutional ethical committee and written informed consent was obtained from all patients.

Patients were not admitted to the study if any of the following criteria were present: (1) patient's refusal, (2) duration of surgery more than 90 minutes, (3) allergy to any drugs of the study, (4) smokers, history of drug or alcohol abuse, (5) treatment with antidepressants, (6) history of diabetes or epilepsy, (7) , history of chronic pain or daily intake of analgesics within 24 h before surgery, (8) treatment with systemic glucocorticoids within 4 weeks before surgery and (9) impaired kidney or liver functions.

Patients were randomly allocated into 3 equal groups, group (I) (GI) (n=25) each patient received Dulox capsule (60mg) orally with sips of water 2 hours preoperatively and 100 ml 0.9% sodium chloride solution (NS) intravenous infusion (IVI) over 15 min (Placebo), group (II) (GII) (n=25) each patient received combined Dulox capsule (60 mg) orally with sips of water and Dex 0.1mg/kg diluted in 100 ml 0.9% NS IVI over 15 min, 2 hours preoperatively and group (III) (GIII) (control group) (n=25) each patient received a placebo capsule identical to Dulox capsule and 100 ml 0.9% NS IVI over 15 min, as a placebo for dexamethasone 2 hours preoperatively. Dulox was presented as CYMBALTA® capsules manufactured by Lilly del Caribe Inc. Imported by Elco and Dex was presented as dexamethasone sulphate ampoules 8mg in 2ml. (Medical Union Pharmaceutical, Egypt MUP). Randomization was done using computer-generated number table of random numbers in a 1:1 ratio and conducted using sequentially numbered, opaque and sealed envelope (SNOSE). Active Dulox capsules were indistinguishable from placebo capsules and placebo capsules contained starch. The study drugs were prepared by the hospital pharmacy and follow-up of patients was conducted by the anesthesia residents not involved in any other part of the study.

During the preoperative anesthetic evaluation, patients were familiarized with 10 cm marked visual analogue scale (VAS) for PO assessment of pain, where 0 cm defines no pain and 10 cm defines the maximum intolerable pain. Patients were also assured that they would receive intramuscular injection (IM) of pethidine 0.5 mg / kg once they experienced pain postoperatively (patients with (VAS > 3).

The general anesthesia technique was standardized for all the patients as well as monitors including 5 lead ECG, non- invasive blood pressure (NIBP) monitor, pulse oximetry and capnography after intubation using Datascope monitors. Neuromuscular function was monitored using a peripheral nerve stimulator. After establishing an intravenous (IV) line, induction of general anesthesia with fentanyl (2 ug/kg) and sleeping dose of propofol followed by rocuronium (0.6 mg/kg) to facilitate orotracheal intubation was done. Anesthesia was maintained using isoflurane in oxygen and air. Ranitidine (50 mg/ampoule) was given diluted in 10 ml 0.9% sodium chloride solution (NS) slowly (IV) over 10 minutes as a gastroprotective regimen. At the end of the surgery, the residual neuromuscular paralysis was antagonized with neostigmine (0.05 mg/kg) and atropine (0.01 mg/kg). After satisfactory recovery, patients were extubated and transferred to the post-anesthesia care unit (PACU) where they were monitored with ECG, NIBP and pulse oximetry.

Assessment of patients' vitals (HR, MAP), arterial SpO2, sedation score, visual analog scale (VAS), the first analgesic requirement time and adverse effects (e.g. nausea, vomiting (PONV), pruritis) were done at 30 minutes, 1h, 2 h, 6h and 12h postoperatively.

PO pain was evaluated at rest based on visual analogue scale, first time to ask for rescue analgesia and total pethidine requirements in 12 hours (mg) postoperatively were recorded. Assessment of sedation was according to sedation score (Ramsay sedation scale) (14).

Hypotension was considered if there was 20% decrease below the baseline for MAP and was treated with IV bolus of ephedrine (3-6 mg). Bradycardia was considered if the heart rate < 55 beats/min and was treated with IV atropine (0.01mg/kg). Respiratory depression was defined as a respiratory rate less than 10 breaths/min-1 or peripheral oxygen saturation less than 95% and was treated with oxygen through a transparent face mask and the intermittent doses of IV naloxone (0.4 mg). IV granisetron (1mg) was given in case of vomiting or after 2 successive episodes of nausea. Pruritus was evaluated with a 4-point scale (0=absent, 1=mild, 2=moderate, 3=severe or requiring treatment), and patients with severe pruritus were treated with IV clemastine (TavegylR) (2 mg / ampoule).

Patient's satisfaction was done by asking the patient to answer the question, 'How would you rate your experience after the surgery?' using a 7-point Likert verbal rating scale (15) and acceptable satisfaction score of the patient being 5-7.

Hormonal stress response was assessed through recording plasma cortisol (micrograms / dl) 2 hours postoperatively. Serum cortisol was measured by a Fluorescence Polarization Immunoassay Technology (FPIA) by the Abbott AXSYM system with the following reference ranges (morning serum cortisol 4.2-38.4 ug/dl) and evening serum cortisol 1.7-16.6 ug/dl).

ELIGIBILITY:
Inclusion Criteria:

female patients aged between 25 and 35 years old of the American Society of Anesthesiologists (ASA) physical status I and II scheduled for elective laparoscopic gynecological surgeries (for infertility) under general anesthesia.

Exclusion Criteria:

1. patient's refusal,
2. duration of surgery more than 90 minutes,
3. allergy to any drugs of the study,
4. smokers, history of drug or alcohol abuse,
5. treatment with antidepressants,
6. history of diabetes or epilepsy,
7. , history of chronic pain or daily intake of analgesics within 24 h before surgery,
8. treatment with systemic glucocorticoids within 4 weeks before surgery and (9) impaired kidney or liver functions. -

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
to compare the analgesic efficacy of Dulox alone, with Dulox and Dex combination in reducing postoperative pain measured by total pethdine requirements 12h after gynecological surgeries. | Total pethdine requirements 12h after gynecological surgeries.